CLINICAL TRIAL: NCT00896168
Title: A Multi-Center, Pre-Marketing Clinical Trial to Evaluate the Efficacy and Safety of Infliximab Treatment on Rheumatoid Arthritis
Brief Title: An Efficacy and Safety Study of Infliximab in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015460; REMICADEART4005
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Infliximab; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab + Methotrexate (Moderate RA) (Experimental): Participants with moderate RA (score greater than 3.2, but less than 5.1 on the disease activity score [DAS] 28) received infliximab 3 milligram per kilogram (mg/kg) intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) at Week 0, 2, 6, 14 and 22 along with oral MTX IN a stable dose of 7.5 to 20 mg per week (equal to the dose used before participation in the study) for 22 weeks.
  Interventions: Drug: Infliximab; Drug: Methotrexate
- Infliximab + Methotrexate (Severe RA) (Experimental): Participants with severe RA (score greater than 5.1 on the DAS 28) received infliximab 3 mg/kg intravenous infusion at Week 0, 2, 6, 14 and 22 along with oral MTX in a stable dose of 7.5 to 20 mg per week (mg/week) equal to the dose used before participation in the study) for 22 weeks.
  Interventions: Drug: Infliximab; Drug: Methotrexate

INTERVENTIONS:
Drug: Infliximab — Infliximab 3 mg per kg intravenous infusion at Week 0, 2, 6, 14 and 22.
Drug: Methotrexate — MTX stable dose (7.5 to 20 mg/week equal to the dose used before participation in the study) for 22 weeks.

SUMMARY:
The purpose of this study is to compare the effectiveness of iInfliximab plus methotrexate (MTX) in treatment of Rheumatoid rheumatoid Arthritis arthritis (RA) (it is an autoimmune disease that causes pain, swelling, stiffness and loss of function in joints) in participants with moderate disease versus participants with severe disease and to compare the efficacy and safety of the MTX subgroups.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (study conducted in more than 1 center), prospective (study following participants forward in time) study comparing the American College of Rheumatology (ACR) scores of participants with moderate RA (defined as having a score greater than 3.2, but less than 5.1 on the Disease Activity Score 28 [DAS 28]) to those participants with severe RA (defined as having a score greater than 5.1 on the DAS 28 score) disease while being treated with infliximab and MTX. DAS evaluates RA activity by several parameters including the number of swollen and tender joints and the participant's own assessment of their pain. Participants will receive infliximab 3 milligram (mg) per kilogram (kg) intravenous infusion (drug given into a vein) (over no less than 2 hours) at Weeks 0, 2, 6, 14 and 22 along oral MTX in a stable dose of 7.5 to 20 mg per week (equal to the dose used before participation in the study) for 22 Weeks. Participants will have a follow-up visit on Week 26. Efficacy will primarily be assessed by the percentage of participants obtaining ACR20, ACR50 and ACR70 response at Week 26. Participants' safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a definitive diagnosis of rheumatoid arthritis (RA) based on the American College of Rheumatology Criteria 1987
* Participants must have been on Methotrexate (MTX) for 12 weeks at the stable dose for at least 4 weeks
* Participants using oral corticosteroids, must have been on a stable dose of prednisone less than 10 milligram per day (mg/day) or its equivalent for at least 4 weeks before screening or if currently not using corticosteroids, the participant must not have received corticosteroids for at least 4 weeks before screening
* Participants with moderate to severe RA (Disease Activity Score [DAS28] greater than 3.2)
* Male participants shall adopt contraceptive measures during the trial and within 6 months after the completion of trial (such as spermicidal barrier), or their female sexual partners shall agree to adopt effective contraceptive measures during the trial or within 6 months after the completion of trial (such as oral contraceptives, contraceptives for injection, intrauterine device [IUD], or sterilization by surgery); female participants of childbearing potential with negative urine pregnancy test upon enrollment in addition to adopting the said contraceptive measures

Exclusion Criteria:

* Participant who has a known allergy to human immunoglobulin proteins or other components of infliximab
* Participant who has a history of receiving infliximab or any other biological preparations
* Participant who is in stage IV RA evaluated by X-ray
* Participants suffering from tuberculosis
* Female participant or male participant's wife who plans to become pregnant during this study and within 6 months after completion of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd. Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab + Methotrexate (Moderate Rheumatoid Arthritis [RA]): Participants with moderate RA (score greater than 3.2, but less than 5.1 on the disease activitiy score [DAS] 28) received infliximab 3 milligram per kilogram (mg/kg) intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) at Week 0, 2, 6, 14 and 22 along oral MTX in a stable dose of 7.5 to 20 mg per week (equal to the dose used before participation in the study) for 22 weeks.
- Infliximab + Methotrexate (Severe RA): Participants with severe RA (score greater than 5.1 on the DAS 28) received infliximab 3 mg/kg intravenous infusion at Week 0, 2, 6, 14 and 22 along with oral MTX in a stable dose of 7.5 to 20 mg per week equal to the dose used before participation in the study) for 22 weeks.
Period: Overall Study
Arm/Group | Infliximab + Methotrexate (Moderate Rheumatoid Arthritis [RA]) | Infliximab + Methotrexate (Severe RA)
Started | 104 | 130
Completed | 90 | 111
Not Completed | 14 | 19
Not completed — Adverse Event | 4 | 7
Not completed — Treatment failure | 8 | 10
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Infliximab + Methotrexate (Moderate RA): Participants with moderate RA (score greater than 3.2, but less than 5.1 on the DAS 28) received infliximab 3 mg/kg intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) at Week 0, 2, 6, 14 and 22 along with oral MTX in a stable dose of 7.5 to 20 mg per week (equal to the dose used before participation in the study) for 22 weeks.
- Total: Total of all reporting groups
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA) | Total
Number analyzed (Participants) | 104 | 130 | 234
Age Continuous [Mean (Standard Deviation); unit: Years] | 42.83 (12.05) | 46.62 (11.39) | 44.92 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 116 | 208
  Male | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology Score 20 Percent (ACR20) Response
Description: ACR20 is achieved if the participant has 20% improvement from Baseline in swollen joint count; tender joint count and in at least 3 of the following 5 assessments: participants' assessment of pain; participants' global assessment of disease activity; physician's global assessment of disease activity; participants' assessment of physical function (Health Assessment Questionnaire [HAQ]) and C-reactive protein (CRP).
Time Frame: Week 26
Population: Full analysis set (FAS) included participants who received at least 1 dose of study medication and had post efficacy data.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Percentage of participants | 63.46 | 76.15

2. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology Score 50 Percent (ACR50) Response
Description: ACR50 is achieved if the participant has 50% improvement from Baseline in swollen joint count; tender joint count and in at least 3 of the following 5 assessments: participants' assessment of pain; participants' global assessment of disease activity; physician's global assessment of disease activity; participants' assessment of physical function (Health Assessment Questionnaire [HAQ]) and C-reactive protein (CRP).
Time Frame: Week 26
Population: The FAS population included participants who received at least 1 dose of study medication and had post efficacy data.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Percentage of participants | 47.12 | 57.69

3. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology Score 70 Percent (ACR70) Response
Description: ACR70 is achieved if the participant has 70% improvement from Baseline in swollen joint count; tender joint count and in at least 3 of the following 5 assessments: participants' assessment of pain; participants' global assessment of disease activity; physician's global assessment of disease activity; participants' assessment of physical function (Health Assessment Questionnaire [HAQ]) and C-reactive protein (CRP).
Time Frame: Week 26
Population: The FAS population included participants who received at least 1 dose of study medication and had post efficacy data.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Percentage of participants | 29.81 | 29.23

4. Secondary Outcome: Change From Baseline in Swollen Joints Count at Week 26
Description: Number of swollen joints were determined by examination of 28 joints and identifying when swelling is present. The number of swollen joints was recorded on the joint assessment form at each visit; the swelling was graded on a scale ranging from 0-2 (0=no swelling, 1=swelling, but bony landmarks seen, 2=swelling but bone marks not seen). Participants categorized as Hepatitis B Virus antigen (HBsAb) positive/negative (at least 1 of HbsAg, HBeAg, Anti-HbeAg and Anti-HbcAg were positive or all were negative).
Time Frame: Baseline and Week 26
Population: The FAS population included participants who received at least 1 dose of study medication and had post efficacy data.
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Swollen joints
  Baseline | 4 (3) | 11 (7)
  Change at Week 26 | -2.6 (3.4) | -7.7 (5.9)

5. Secondary Outcome: Change From Baseline in Tender Joints Count at Week 26
Description: Number of tender joints was determined by examination of 28 joints and identifying when tenderness is present. The number of tender joints was recorded on the joint assessment form at each visit; the tenderness of symptomatic joints was graded on a scale ranging from 0-3 (0=no pain, 1=mild, 2= moderate and 3=severe).
Time Frame: Baseline and Week 26
Population: The FAS population included participants who received at least 1 dose of study medication and had post efficacy data.
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Tender joints
  Baseline | 6 (4) | 15 (8)
  Change at Week 26 | -4.0 (4.1) | -10.6 (8.0)

6. Secondary Outcome: Change From Baseline in Participant's Pain Visual Analogue Scale (VAS) Score at Week 26
Description: Participant's pain was assessed on VAS of 0 to 100 mm (0=not at all to 100=extreme pain).
Time Frame: Baseline and Week 26
Population: The FAS population included participants who received at least 1 dose of study medication and had post efficacy data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Units on a scale
  Baseline | 47 (16) | 67 (18)
  Change at Week 26 | -26.8 (21.9) | -37.3 (27.9)

7. Secondary Outcome: Change From Baseline in Participants' Global Disease Assessment at Week 26
Description: Participants scored the overall disease state using VAS of 0-100 mm. Participants might have assessed the Control of their current disease using "0 mm=very good" to "100 mm=very poor" scale.
Time Frame: Baseline and Week 26
Population: The FAS population included participants who received at least 1 dose of study medication and had post efficacy data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Units on a scale
  Baseline | 49 (17) | 68 (17)
  Change at Week 26 | -28.3 (23.3) | -39.3 (27.1)

8. Secondary Outcome: Change From Baseline in Physicians' Global Disease Assessment at Week 26
Description: Physicians scored the overall disease state using VAS of 0-100 mm. Physicians might have assessed the activity of RA using "0=no active RA" to "100=most serious active RA" scale.
Time Frame: Baseline and Week 26
Population: FAS population included participants who received at least 1 dose of study medication and possessed the record of efficacy data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Units on a scale
  Baseline | 46 (17) | 67 (18)
  Change at Week 26 | -25.3 (21.7) | -36.4 (23.1)

9. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 26
Description: Duration of morning stiffness: Time elapsed in minutes when participant woke up in morning and was able to resume normal activities without stiffness. Increase in stiffness duration from Baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Minutes
  Baseline | 44.73 (61.97) | 102.58 (144.36)
  Change at Week 26 | -36.63 (68.38) | -77.12 (84.73)

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) at Week 26
Description: The HAQ, a 20-question instrument, assesses the degree of difficulty a person has in accomplishing tasks in eight functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores). Responses in each area are scored from 0=no difficulty to 3=inability to perform a task in that area.
Time Frame: Baseline and Week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Units on a scale
  Baseline | 0.9 (0.6) | 1.3 (0.8)
  Change at Week 26 | -0.59 (0.58) | -0.83 (0.67)

11. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 26
Description: CRP is a protein found in the blood, the levels of which rise in response to inflammation.
Time Frame: Baseline and Week 26
Population: FAS population included participants who received at least 1 dose of study medication and possessed the record of efficacy data. Here, 'N' signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Milligram/Liter
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 103 | 128
Milligram/Liter
  Baseline | 1.24 (1.71) | 2.93 (4.26)
  Change at Week 26 | -0.54 (1.52) | -1.22 (4.69)

12. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 26
Description: ESR is also called a sedimentation rate or Westergren ESR, is the rate at which red blood cells sediment in a period of 1 hour. It is a common hematology test, and is a non-specific measure of inflammation.
Time Frame: Baseline and Week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeter/1 hour
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Number analyzed (Participants) | 104 | 130
Millimeter/1 hour
  Baseline | 24.45 (16.62) | 51.34 (28.66)
  Change at Week 26 | -2.19 (17.82) | -16.53 (29.77)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Arm/Group | Infliximab + Methotrexate (Moderate RA) | Infliximab + Methotrexate (Severe RA)
Serious Adverse Events (participants affected / at risk) | 2/104 | 2/130
Other Adverse Events (participants affected / at risk) | 57/104 | 80/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab + Methotrexate (Moderate RA) (N=104) | Infliximab + Methotrexate (Severe RA) (N=130)
Tuberculosis (Immune system disorders) | 0 | 1
Fungal pneumonia (Immune system disorders) | 0 | 1
Septicemia (Immune system disorders) | 1 | 0
Cardiac disorders (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab + Methotrexate (Moderate RA) (N=104) | Infliximab + Methotrexate (Severe RA) (N=130)
Hypertension (Cardiac disorders) | 4 | 3
Hypolekocytosis (Blood and lymphatic system disorders) | 4 | 14
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 29 | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Hepatic function disnormal (Hepatobiliary disorders) | 52 | 49
Nausea (Gastrointestinal disorders) | 4 | 4
Skin rash (Skin and subcutaneous tissue disorders) | 1 | 13
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Fever (General disorders) | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days